CLINICAL TRIAL: NCT03763149
Title: A Phase 1a Study Evaluating the Safety, Tolerability, and Initial Efficacy of Recombinant Human Anti-cluster Differentiation Antigen 47 (CD47) Monoclonal Antibody Injection (IBI188) in Patients With Advanced Malignant Tumors and Lymphomas
Brief Title: A Study Evaluating the Safety, Tolerability, and Initial Efficacy of Recombinant Human Anti-cluster Differentiation Antigen 47 (CD47) Monoclonal Antibody Injection (IBI188) in Patients With Advanced Malignant Tumors and Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI188A102
Record Dates: First submitted 2018-11-18; First posted 2018-12-04 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IBI188 (Experimental): Part 1: Accelerated Titration Phase 0.1 mg/kg IV; QW 0.3 mg/kg IV QW; 1 mg/kg IV QW
  Part 2 : Dose Escalation Phase with initial fixed priming dose Priming dose of 1mg/kg on C1D1 followed by 3 mg/kg IV QW; 10 mg/kg IV QW; 20 mg/kg IV QW; 30 mg/kg IV QW.
  Interventions: Biological: IBI188

INTERVENTIONS:
Biological: IBI188 — The study is composed of two stages: Part 1 Accelerated Titration Phase and Part 2 Dose Escalation Phase with initial fixed priming dose.
  The starting dose for part 1 is 0.1 mg/kg QW, followed by 2 dose cohorts (0.3 mg/kg QW and 1 mg/kg QW). Duration of dose limiting toxicity (DLT) observation is 28 days.
  Part 2 will have 4 dose cohorts(3mg/kg QW、10mg/kg QW、20mg/kg QW and 30mg/kg QW). Conventional 3+3 Dose Escalation will be adopted. DLT observation period is 28 days.

SUMMARY:
This is an open-label, dose escalation, Phase I study to evaluate the safety, tolerability, pharmacokinetics and efficacy in patients with advanced malignancies.

DETAILED DESCRIPTION:
The study is composed of two stages: Part 1 Accelerated Titration Phase and Part 2 Dose Escalation Phase with initial fixed priming dose.

The starting dose for part 1 is 0.1 mg/kg QW, followed by 2 dose cohorts (0.3 mg/kg QW and 1 mg/kg QW). Duration of dose limiting toxicity (DLT) observation is 28 days.

Part 2 will have 4 dose cohorts(3mg/kg QW、10mg/kg QW、20mg/kg QW and 30mg/kg QW). Conventional 3+3 Dose Escalation will be adopted. DLT observation period is 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the ICF.
2. Male or female subject above18 years.
3. Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumors and lymphomas that are refractory to standard therapy, or for which no standard therapy exists.
4. For dose expansion at the RP2D: subject has measurable disease per RECIST v1.1. that was not in a prior radiation area within past 6 months, unless tumor growth was documented following radiation. Lymphomas have at least one measurable lesion and FDG-avid lesion according to the Lugano 2014 criteria.
5. Separate informed consent for subjects who provide archived tissue biopsies for biomarker testing (Optional).
6. ECOG Performance Status 0 to 1
7. Subjects with life expectancy of ≥ 3 month
8. No herbal/alternative medications within 14 days prior to the first dose of IBI188.
9. Must have adequate organ function, prior to start of IBI188, including the following:

   1. Bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.5 x109/L; platelet count ≥ 100 x 109/L; hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L; Lymphocyte counts ≥ 0.5 x109/L
   2. Hepatic: total bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 X ULN (≤5 X ULN if with liver involvement)
   3. Renal: serum creatinine ≤ 1.5 times the ULN or estimated creatinine clearance ≥50mL/min (Cockroft and Gault formula [https://www.mdcalc.com/creatinine-clearance-cockcroft-gault-equation]).
   4. Coagulation tests INR < 2.0, activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
10. Subjects (women of child-bearing potential and males) must be willing to use viable contraception method that is deemed effective by the investigator throughout the treatment period and for at least three months following the last dose of study drug. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:

1. Pregnant or nursing females.
2. Any remaining AEs > grade 1 from prior anti-tumor treatment as per CTCAE v5.0, with exception of the residual hair loss;
3. Received a biologic G-CSF, GM-CSF or erythropoietin within 14 days prior to the first dose of study drug;
4. Subjects participating in any other interventional clinical study
5. Previous exposure to any anti-CD47 monoclonal antibody or SIRPα antibody.
6. Subjects who had transfusion within 3 weeks
7. Patients who are on anticoagulants and /or require concomitant aspirin or other nonsteroidal anti-inflammatory medications.
8. Subjects who have a history of documented autoimmune disease, even if not clinically severe or never treated with systemic steroids or immunosuppressive agents, are not candidates for this clinical trial, except for autoimmune hypothyroidism and well-controlled Type 1 diabetes mellitus.
9. Subjects with or w/o autoimmune condition requiring systemic treatment with either corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive medications within 14 days before the planned first dose of study drug. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease. Ophthalmologic, nasal and intra-articular injections or steroids are acceptable.
10. Subject with primacy central nervous system (CNS) malignancy or symptomatic CNS metastases are not allowed. Subjects with asymptomatic CNS metastases are eligible if clinically controlled, which is defined as ≥8 weeks of stable neurologic function following CNS-directed therapy, and no evidence of CNS disease progression as determined by radiographic imaging ≥ 4 weeks prior to screening. No interim progression between the completion of CNS-directed therapy and the screening tumor assessment, and ≥ 2 weeks from discontinuation of anti-seizure and steroid therapies from screening.
11. Subjects who have had major surgery within the 28-days from the screening;
12. Subjects with idiopathic pulmonary fibrosis or unresolved active or chronic inflammatory pulmonary disease are excluded. Subjects with a history of radiation pneumonitis which has resolved are eligible.
13. Positive for human immunodeficiency virus (HIV) infection.
14. Active hepatitis B or C. HBV carriers without active disease (HBV DNA titer< 1000 cps/mL or 200 IU/mL), or cured Hepatitis C (negative HCV RNA test) may be enrolled.
15. History of primary immunodeficiency, stem cell or organ transplant, or previous clinical diagnosis of tuberculosis disease.
16. Subject who have had severe infection deemed clinically significant per investigator within 4 weeks or signs and symptoms of any active infection within 2 weeks prior to the first dose administration.
17. Known allergies, hypersensitivity, or intolerance to protein-based therapies or with a history of any significant drug allergy (e.g., anaphylaxis, hepatotoxicity, immune-mediated thrombocytopenia or anemia).
18. Subjects who experienced immunotherapy-related adverse events (irAE) grade ≥ 3, or who had to discontinue prior immunotherapy treatment due to irAEs of any grade.
19. Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure (New York Heart Association) NYHA III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 6 months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
20. Any other serious underlying medical (e.g. uncontrolled diabetes mellitus, uncontrolled hypertension, active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect subject compliance or place the subject at high risk from treatment-related complications.
21. Known history of hypersensitivity to any components of the IBI188 product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Number of patients with AEs and SAEs | 2 years
  To evaluate the safety and tolerability of IBI188 [Adverse events (AEs), Serious Adverse Events (SAE) ]

SECONDARY OUTCOMES:
Pharmacokinetics: AUC | up to 2 years after enrollment
  The area under the curve (AUC) of serum concentration of the drug after the administration
Pharmacokinetics: Cmax | up to 2 years after enrollment
  Maximum concentration(Cmax) of the drug after administration
Immunogenicity: Percentage of ADA positive patients | up to 2 years after enrollment
  Number of Anti-Drug Antibodies (ADA) positive patients will be counted and percentage of ADA positive patients will be calculated to evaluate immunogenicity of IBI188.
Preliminary anti-tumor activity of IBI188 (Objective Response Rate) | up to 2 years after enrollment
  Objective Response Rate (ORR) is the percentage of Complete Response (CR) plus partial response (PR) assessed by iRECIST v1.1 criteria for solid tumors and Lugano2014 criteria for lymphoma.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - START Midwest, Grand Rapids, Michigan
  - Thomas Jefferson Univerity, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - START (South Texas Accelerated Research Therapeutics, LLC), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No